CLINICAL TRIAL: NCT00414557
Title: The Effects of Knee Malalignment and Quadriceps Strengthening on the Adduction Moment in Individuals With Medial Knee Osteoarthritis
Brief Title: Knee Malalignment and Thigh Muscle Strengthening in Individuals With Medial Knee Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Australian Physiotherapy Research Foundation (Other); United Pacific Industries (Unknown)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 040850
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2006-12-22 (Estimated); Status verified 2006-12

CONDITIONS: Knee Osteoarthritis
Keywords: Musculoskeletal diseases; Joint diseases
MeSH Terms: conditions — Osteoarthritis, Knee; Musculoskeletal Diseases; Joint Diseases

INTERVENTIONS:
Procedure: Quadriceps strengthening

SUMMARY:
To investigate the effects of quadriceps strengthening on the adductor moment in individuals with medial knee OA and whether quadriceps strengthening has a different effect on the adductor moment in individuals with and without knee malalignment

DETAILED DESCRIPTION:
Although quadriceps strengthening is the cornerstone of physiotherapy management, recent evidence suggests that high quadriceps strength in patients with malaligned knees may increase OA progression.

This study investigates the effects of quadriceps strengthening on the adduction moment in patients with medial knee OA with and without malalignment. 107 participants with and without varus knee malalignment were recruited and randomised into an exercise or a control group. Participants in the exercise group were taught five quadriceps strengthening exercises by a project physiotherapist to be performed five days a week for twelve weeks at home. The exercises were:

1. Quadriceps exercise over fulcrum using ankle weight
2. Straight leg raise exercise using ankle weight
3. Long arc knee extension exercise in sitting using ankle weight
4. Knee extension exercise with isometric hold at 60° knee flexion using ankle weight
5. Knee extension exercise with isometric hold at 60° knee flexion using an elastic band.

Each exercise was performed at 2x10 repetitions for the first 2 weeks and 3x10 repetitions thereafter.

Participants visited the physiotherapist 7 times at Week 1, 2, 3, 4, 5, 7 and 10. They were given the ankle weights and elastic band to bring home and instructed about the repetitions and weights to use by the physiotherapist, who also checked and progressed their exercises. The average duration of the physiotherapy sessions was 30 minutes. To monitor compliance, each participant was given an exercise instructions sheet and kept a training diary to record the exercises they had done.

The control group received no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pain in the knee
* Osteophytes on knee x-ray
* Self-reported pain on the inner aspect of the study knee
* Osteophytes in the medial compartment of the knee joint and
* Medial joint space narrowing greater than lateral joint space narrowing on x-ray

Exclusion Criteria:

* Knee surgery within the previous 6 months
* History of lower limb joint replacements
* Systemic arthritic conditions such as rheumatic or psoriatic arthritis
* Valgus knee deformity (> 5º)
* Inability to walk without the use of walking aids
* Intending to start a lower limb strengthening program in the next 3 months
* Seeking or currently receiving physiotherapy for OA knee

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107
Dates: Start 2004-05; Study Completion 2006-12

PRIMARY OUTCOMES:
Adduction moment
Time points: 0 and 13 weeks

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire
Numerical rating scales for pain
Quadriceps and hamstrings strength
Self-selected walking speed
Dynamic balance using step test
Physical function using stair climb test
Time points: 0 and 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kim Bennell, PhD, Principal Investigator — University of Melbourne; Rana Hinman, PhD, Principal Investigator — University of Melbourne; Tim Wrigley, MSc, Principal Investigator — University of Melbourne; Boon W Lim, MSc, Principal Investigator — University of Melbourne; Leena Sharma, MD, Principal Investigator — Northwestern University Medical School, Chicago
Locations (1):
- The University of Melbourne, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Lim BW, Hinman RS, Wrigley TV, Sharma L, Bennell KL. Does knee malalignment mediate the effects of quadriceps strengthening on knee adduction moment, pain, and function in medial knee osteoarthritis? A randomized controlled trial. Arthritis Rheum. 2008 Jul 15;59(7):943-51. doi: 10.1002/art.23823. PMID 18576289